CLINICAL TRIAL: NCT03749785
Title: The Effect of Carbohydrate Feeding Frequency on Muscle Glycogen and Exercise Capacity in Runners
Brief Title: Carbohydrate Feeding Frequency, Muscle Glycogen and Exercise Capacity in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Betts, Professor, Department for Health, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18/SW/0177
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular carbohydrate feeding (Active Comparator): Ingestion of 75 g sucrose, given in regular doses for the first 75 minutes of exercise during a time to exhaustion run
  Interventions: Other: Regular carbohydrate feeding
- Single carbohydrate bolus (Active Comparator): Ingestion of 75 g sucrose, given in a single bolus after 75 minutes of exercise, during a time to exhaustion run
  Interventions: Other: Single carbohydrate bolus

INTERVENTIONS:
Other: Regular carbohydrate feeding — 60 ml of water with 5 g sucrose given every 5 minutes 14 times up until 70 minutes followed by 5 g sucrose after 75 minutes in a 250 ml solution
  Arms: Regular carbohydrate feeding
Other: Single carbohydrate bolus — 60 ml of water given every 5 minutes 14 times up until 70 minutes followed by 75 g sucrose after 75 minutes in a 250 ml solution
  Arms: Single carbohydrate bolus

SUMMARY:
The aim of this study is to investigate the effects of regular sucrose feeds compared to a single large bolus given late in exercise, on muscle glycogen utilisation, exercise capacity and other markers of metabolism during running

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a trained runner
* Regularly participate in running activity (>2 times a week)
* Participated in running based training for a minimum of 2 years
* Be willing to undertake exercise sessions until volitional exhaustion
* Be willing to have the necessary samples taken during the testing protocols
* Not a habitual smoker
* Have the capacity and willingness to provide informed consent (oral and written)
* Successful completion of the physical activity readiness questionnaire (PAR-Q)

Exclusion Criteria:

* Female
* <18 or >50 years old
* Not regularly participating in running activity (<3 times a week)
* Experience contraindications to the administration of the proposed anaesthetic (Lidocaine Hydrochloride)
* Habitual/previously habitual smoker

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Muscle glycogen concentrations | Estimated to be between 90 and 145 minutes
  Muscle glycogen concentration at rest, after 75 minutes of treadmill running and at volitional exhaustion. Measured using the bergstrom needle technique for obtaining muscle biopsy samples
Exercise capacity | Estimated to be between 90 and 145 minutes
  Time to exhaustion at the pre-determined speed to elicit exhaustion after ~90 minutes when ingesting water only

SECONDARY OUTCOMES:
Ratings of perceived exertion | Estimated to be between 90 and 145 minutes
  Subjective ratings of perceived exertion, during treadmill running. Measured using a borg scale of 6 to 20, where 6 = no exertion at all, and 20 = maximal exertion.
Ratings of stomach discomfort | Estimated to be between 90 and 145 minutes
  Subjective ratings of stomach discomfort during treadmill running. Measured using a modified borg scale of 6 to 20, where 6 = no discomfort and 20 = maximal discomfort
Carbohydrate oxidation | Estimated to be between 90 and 145 minutes
  Total carbohydrate oxidation during treadmill running. Measured using indirect calorimetry and reported in grams.
Fat oxidation | Estimated to be between 90 and 145 minutes
  Total fat oxidation during treadmill running. Measured using indirect calorimetry and reported in grams.
Plasma glucose concentrations | Estimated to be between 90 and 145 minutes
  Plasma lactate concentrations during of treadmill running. Measured using colourimetric assay and reported in mmol/L
Plasma lactate concentrations | Estimated to be between 90 and 145 minutes
  Plasma lactate concentrations during treadmill running. Measured using colourimetric assay and reported in mmol/L.
Heart rate | Estimated to be between 90 and 145 minutes
  Heart rate during treadmill running measured by telemetry and reported in beats per minute
Rate of oxygen consumption | Estimated to be between 90 and 145 minutes
  Rate of oxygen consumption during treadmill running. Measured using indirect calorimetry and reported in litres per minute
Rate of carbon dioxide production | Estimated to be between 90 and 145 minutes
  Rate of carbon dioxide production during treadmill running. Measured using indirect calorimetry and reported in litres per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom